CLINICAL TRIAL: NCT04456712
Title: Effect of Ciprofloxacin Versus Levofloxacin on QTc-interval and Dysglycemia in Diabetic and Non-Diabetic Patients.
Brief Title: Effect of Ciprofloxacin Versus Levofloxacin on QTc-interval and Dysglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nada Abd El-Hamed Saad Rezk, clinical pharmacist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ciprofloxacin and levofloxacin
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: QTc Prolongation, Hyperglycemia, Hypoglycemia
Keywords: Levofloxacin, ciprofloxacin, QTc prolongation, dysglycemia.
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia | interventions — Ciprofloxacin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: fifty diabetic patients received intravenous levofloxacin 750 mg/24 hours. fifty diabetic patients received intravenous ciprofloxacin 400mg/12 hours. fifty non-diabetic patients received intravenous levofloxacin 750 mg/24 hours. fifty non-diabetic patients received intravenous ciprofloxacin 400mg/12 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ciprofloxacin for diabetic patients (Experimental): 50 diabetic patients received intravenous ciprofloxacin 400mg/12 hours.
  Interventions: Drug: Ciprofloxacin 400 MG/200 ML Intravenous Solution
- levofloxacin for diabetic patients (Experimental): 50 diabetic patients received intravenous levofloxacin 750mg/24 hours.
  Interventions: Drug: Levofloxacin 750 MG
- ciprofloxacin for non-diabetic patients (Experimental): 50 non-diabetic patients received intravenous ciprofloxacin 400mg/12 hours.
  Interventions: Drug: Ciprofloxacin 400 MG/200 ML Intravenous Solution
- levofloxacin for non-diabetic patients (Experimental): 50 non-diabetic patients received intravenous levofloxacin 750mg/24 hours.
  Interventions: Drug: Levofloxacin 750 MG

INTERVENTIONS:
Drug: Ciprofloxacin 400 MG/200 ML Intravenous Solution — antibiotic
  Arms: ciprofloxacin for diabetic patients; ciprofloxacin for non-diabetic patients
Drug: Levofloxacin 750 MG — antibiotic
  Arms: levofloxacin for diabetic patients; levofloxacin for non-diabetic patients

SUMMARY:
To compare intravenous levofloxacin and ciprofloxacin regarding their risk on the corrected QT interval (QTc) prolongation and dysglycemia in diabetic and non-diabetic patients.

DETAILED DESCRIPTION:
Fluoroquinolones represent an important class of antibacterial drug and they are used worldwide.Fluoroquinolones are classified into generations according to the spectrum of antimicrobial activities that targeted them.Fluoroquinolones may cause several side effects as tendon rupture, central nervous toxicity, cardiovascular toxicity, gastrointestinal toxicity, phototoxicity, disrupted glucose metabolism, skin disorders and hypersensitivity. Ciprofloxacin, a second generation fluoroquinolone, is one of the most successful and widely used compounds of fluoroquinolone. On the other hand, levofloxacin is a third generation fluoroquinolone.

Diabetes mellitus (DM) is chronic disease and a serious of metabolic disorder associated with the presence of hyperglycemia due to partial or complete insulin deficiency. Diabetes mellitus is a major risk factor for cardiovascular diseases.

Fluoroquinolone class is associated with cardiac side effects as QTc prolongation. Some agents of fluoroquinolones were withdrawn from market. However, cardiac adverse effects has been developed with fluoroquinolones still in market. Members of fluoroquinolones class have different effects on QT interval. The US FDA suggested that the risk and benefits ratio of fluoroquinolones should be taken into consideration.

In addition to hyperglycemia events are more common with fluoroquinolones than with other classes of antibiotics. The food and drug administration (FDA) confirmed the current warning that fluoroquinolones may cause decrease in blood sugar especially in diabetic patients. However, other study proved that fluoroquinolones may cause dysglycemic events in diabetic and non-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (male, female)
* age from 18 to 70 years .
* Be able to give an informed consent form after understanding for reasonable explanation of clinical trial's purpose, contents and characteristics of clinical drugs
* Wiling to participate whole clinical trial periods

Exclusion Criteria:

* Younger than 18 years or older than 70 years.
* Has prolonged QTc before receiving therapy.
* With a history of heart diseases.
* Received class IA or III antiarrhythmic agents.
* Received macrolide antibiotics.
* With a history of quinolone allergy.
* Pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Effect of ciprofloxacin versus levofloxacin on QTc interval | before starting antibiotic, after 24 hours, 72 hours from the first dose and after 72 hours from antibiotic cessation
  change in QTc interval (QTc prolongation)
Effect of ciprofloxacin versus levofloxacin on fasting blood glucose | before starting antibiotic, after 24 hours, 72 hours from the first dose and after 72 hours from antibiotic cessation
  change in fasting blood glucose (dysglycemia)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Elberry, professor, Study Director — Faculty of medicine, Beni-Suef university, Beni-Suef, Egypt; Hazem S Hussein, MD, Study Director — Faculty of medicine, Beni-Suef university, Beni-Suef, Egypt; Raghda R Sayed, PhD, Study Director — Faculty of pharmacy, Beni-Suef university, Beni-Suef, Egypt
Locations (1):
- Beni-Suef university hospital, Cairo, Egypt

REFERENCES:
- [Background] Mathews B, Thalody AA, Miraj SS, Kunhikatta V, Rao M, Saravu K. Adverse Effects of Fluoroquinolones: A Retrospective Cohort Study in a South Indian Tertiary Healthcare Facility. Antibiotics (Basel). 2019 Jul 27;8(3):104. doi: 10.3390/antibiotics8030104. PMID 31357640
- [Background] Lu ZK, Yuan J, Li M, Sutton SS, Rao GA, Jacob S, Bennett CL. Cardiac risks associated with antibiotics: azithromycin and levofloxacin. Expert Opin Drug Saf. 2015 Feb;14(2):295-303. doi: 10.1517/14740338.2015.989210. Epub 2014 Dec 10. PMID 25494485
- [Background] Granados J, Ceballos M, Amariles P. [Hypo or hyperglycemia associated with fluoroquinolone use]. Rev Med Chil. 2018 May;146(5):618-626. doi: 10.4067/s0034-98872018000500618. Spanish. PMID 30148925
- [Background] Gonzalez M C, Rosales C R, Pavez D, Fuenzalida LM, Soto A, Perez R, Perez J, Araos R, Pinto ME. [Safety of fluoroquinolones: risks usually forgotten for the clinician]. Rev Chilena Infectol. 2017 Dec;34(6):577-582. doi: 10.4067/S0716-10182017000600577. Spanish. PMID 29488552